CLINICAL TRIAL: NCT06783049
Title: Secondary Prevention of Ischemic Stroke and Transient Ischemic Attack With an Intelligent System
Brief Title: Secondary Prevention of Ischemic Stroke and Transient Ischemic Attack With an Intelligent Management System
Acronym: SPIRIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Tsinghua Chang Gung Hospital (Other); Xiangya Hospital of Zhongnan University (Unknown); The affiliated Hospital of Shihezi University (Unknown); The First Hospital of Jilin University (Other); First People's Hospital of Foshan (Other); The Second Affiliated Hospital of Fujian Medical University (Other); BOE Technology Group Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Zi-Xiao Li, Principal Investigator, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022YFC250494
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack (TIA)
Keywords: ischemic stroke; secondary prevention; digital health
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in the control group received secondary stroke prevention discharge recommendations from their attending physicians, based on standard medical practice. No additional interventions for secondary prevention were applied throughout the study.
- Intervention group (Experimental)
  Interventions: Behavioral: Cerebrovascular Disease Secondary Prevention Smart Management System

INTERVENTIONS:
Behavioral: Cerebrovascular Disease Secondary Prevention Smart Management System — The continuous post-discharge intervention for patients was conducted using the Cerebrovascular Disease Secondary Prevention Smart Management System. This system, integrated with a WeChat-based applet, records patients' basic information and connects with mobile IoT devices such as blood pressure monitors and glucose meters. This allows patients to self-monitor their risk factors post-discharge. Based on international guidelines, high-level evidence, and the clinical expertise of cerebrovascular specialists, a comprehensive clinical decision-making tree was developed. This serves as the foundation for an AI feedback system that provides intelligent feedback on risk factor control and predicts the risk of recurrence.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to develop a digital health-based intelligent management system for the secondary prevention of ischemic stroke and to evaluate its effectiveness through a multicenter randomized controlled trial, assessing its health economic value.

Participants will receive usual care after discharge (control group) or be managed with a WeChat-based intelligent management system after discharge (intervention group).

At one year, all patients will undergo face-to-face follow-up to assess clinical events, medication adherence, and the achievement of target risk factor levels.

DETAILED DESCRIPTION:
Before discharge, patients receive standard education on the secondary prevention of ischemic stroke from their physician, covering topics such as secondary prevention medications, risk factor management, lifestyle modifications, and rehabilitation. Additionally, the "Intelligent Management System," a WeChat-based applet, is activated for each patient. The system records basic patient information and integrates with mobile IoT devices, such as blood pressure monitors and glucose meters, allowing for self-monitoring of risk factors post-discharge. Based on international guidelines, high-level evidence, and the expertise of stroke specialists, a comprehensive clinical decision-making tree is established. This serves as the foundation for an AI feedback system that provides intelligent feedback on risk factor control and predicts recurrence risk. The patient interface includes educational content on ischemic stroke, risk factor management, lifestyle adjustments, and follow-up schedules post-discharge.

The system also features a physician interface, which enables attending doctors to offer online consultations, schedule face-to-face follow-up appointments, and manage patients long-term. Each patient is assigned to an "Online Stroke Care Team," which includes a "Health Management Officer" responsible for facilitating communication between the patient and the physician and providing basic health guidance. Additionally, an "Online Doctor" is available to answer stroke-related medical questions.

The Health Management Officer monitors patients' health data and arranges online or in-person consultations for those with poor adherence or suboptimal target achievement. Patient management is guided by the theory of health empowerment, creating an integrated online and offline ischemic stroke management intervention model.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients diagnosed with acute ischemic stroke or transient ischemic attack.
3. Time from onset to enrollment ≤ 14 days.
4. Presence of at least one modifiable risk factor (hypertension, diabetes).
5. Ability to independently use a smartphone to complete system tasks upon discharge, or with the assistance of family members.
6. Signed informed consent by the patient or their family members.

Exclusion Criteria:

1. Patients already enrolled in other stroke-related healthcare quality improvement projects or clinical trials.
2. Patients or family members who refuse to sign the informed consent form.
3. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4490 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Vascular events and all-causes death | From enrollment to 1 year follow-up
  Vascular and all-cause mortality events were collected for one year post-enrollment through face-to-face follow-ups and patient self-reports. Vascular events included stroke recurrence, transient ischemic attacks, myocardial infarction, vascular interventions or surgeries, and systemic embolism. If a patient experienced both a vascular event and death, only one event was recorded. In cases of multiple vascular events, only the first event was documented.
Risk factor control rate | From enrollment to 1 year follow-up
  Risk factor control was defined as achieving glycated hemoglobin (HbA1c) ≤7% or blood pressure below the target set at discharge. If a patient had both hypertension and diabetes at enrollment, meeting the criteria for both conditions was considered two achieved targets. If the patient had only hypertension or diabetes at enrollment, meeting the target for the respective condition was considered one achieved target.

SECONDARY OUTCOMES:
Readmission to hospital within 1 year | From enrollment to 1 year follow-up
Stroke-related readmission | From enrollment to 1 year follow-up
Direct medical costs | From enrollment to 1 year follow-up
Rate of good adherence to secondary prevention medicine | From enrollment to 1 year follow-up
Adverse drug reaction | From enrollment to 1 year follow-up
Body mass index | From enrollment to 1 year follow-up
Waist circumstance | From enrollment to 1 year follow-up
Frequency of blood pressure monitoring | From enrollment to 1 year follow-up
  calculated as time/week
Frequency of blood glucose monitoring | From enrollment to 1 year follow-up
  calculated as time/week
Blood lipid levels | From enrollment to 1 year follow-up
  Included total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglyceridee
Rehabilitation | From enrollment to 1 year follow-up
Smoking | From enrollment to 1 year follow-up
Alcohol | From enrollment to 1 year follow-up
Regular exercise | From enrollment to 1 year follow-up
Overall physical activity level | From enrollment to 1 year follow-up
  Assessed by IPAQ-S, calculated as MET-min/week
Fatigue | From enrollment to 1 year follow-up
  Assessed by Fatigue Severity Scale (FSS). Fatigue was defined as total FSS score ≥36

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang
  - Beijing Tiantan Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonura A, Motolese F, Capone F, Iaccarino G, Alessiani M, Ferrante M, Calandrelli R, Di Lazzaro V, Pilato F. Smartphone App in Stroke Management: A Narrative Updated Review. J Stroke. 2022 Sep;24(3):323-334. doi: 10.5853/jos.2022.01410. Epub 2022 Sep 30. PMID 36221935
- [Result] Schwamm LH. Digital Health Strategies to Improve Care and Continuity Within Stroke Systems of Care in the United States. Circulation. 2019 Jan 8;139(2):149-151. doi: 10.1161/CIRCULATIONAHA.117.029234. No abstract available. PMID 30615498
- [Result] Requena M, Montiel E, Baladas M, Muchada M, Boned S, Lopez R, Rodriguez-Villatoro N, Juega J, Garcia-Tornel A, Rodriguez-Luna D, Pagola J, Rubiera M, Molina CA, Ribo M. Farmalarm. Stroke. 2019 Jul;50(7):1819-1824. doi: 10.1161/STROKEAHA.118.024355. Epub 2019 Jun 6. PMID 31167621
- [Result] Kim BJ, Park JM, Park TH, Kim J, Lee J, Lee KJ, Lee J, Chae JE, Thabane L, Lee J, Bae HJ. Remote blood pressure monitoring and behavioral intensification for stroke: A randomized controlled feasibility trial. PLoS One. 2020 Mar 11;15(3):e0229483. doi: 10.1371/journal.pone.0229483. eCollection 2020. PMID 32160205
- [Result] Allan LP, Beilei L, Cameron J, Olaiya MT, Silvera-Tawil D, Adcock AK, English C, Gall SL, Cadilhac DA. A Scoping Review of mHealth Interventions for Secondary Prevention of Stroke: Implications for Policy and Practice. Stroke. 2023 Nov;54(11):2935-2945. doi: 10.1161/STROKEAHA.123.043794. Epub 2023 Oct 6. PMID 37800373
- [Result] Ahmadi M, Laumeier I, Ihl T, Steinicke M, Ferse C, Endres M, Grau A, Hastrup S, Poppert H, Palm F, Schoene M, Seifert CL, Kandil FI, Weber JE, von Weitzel-Mudersbach P, Wimmer MLJ, Algra A, Amarenco P, Greving JP, Busse O, Kohler F, Marx P, Audebert HJ. A support programme for secondary prevention in patients with transient ischaemic attack and minor stroke (INSPiRE-TMS): an open-label, randomised controlled trial. Lancet Neurol. 2020 Jan;19(1):49-60. doi: 10.1016/S1474-4422(19)30369-2. Epub 2019 Nov 7. PMID 31708447
- [Result] Duncan PW, Bushnell CD, Jones SB, Psioda MA, Gesell SB, D'Agostino RB Jr, Sissine ME, Coleman SW, Johnson AM, Barton-Percival BF, Prvu-Bettger J, Calhoun AG, Cummings DM, Freburger JK, Halladay JR, Kucharska-Newton AM, Lundy-Lamm G, Lutz BJ, Mettam LH, Pastva AM, Xenakis JG, Ambrosius WT, Radman MD, Vetter B, Rosamond WD; COMPASS Site Investigators and Teams.. Randomized Pragmatic Trial of Stroke Transitional Care: The COMPASS Study. Circ Cardiovasc Qual Outcomes. 2020 Jun;13(6):e006285. doi: 10.1161/CIRCOUTCOMES.119.006285. Epub 2020 Jun 1. PMID 32475159
- [Result] Ihl T, Ahmadi M, Laumeier I, Steinicke M, Ferse C, Klyscz P, Endres M, Hastrup S, Poppert H, Palm F, Kandil FI, Weber JE, von Weitzel-Mudersbach P, Wimmer MLJ, Audebert HJ. Patient-Centered Outcomes in a Randomized Trial Investigating a Multimodal Prevention Program After Transient Ischemic Attack or Minor Stroke: The INSPiRE-TMS Trial. Stroke. 2022 Sep;53(9):2730-2738. doi: 10.1161/STROKEAHA.120.037503. Epub 2022 Jun 15. PMID 35703097
- [Result] Song J, Wang X, Wang B, Ge Y, Bi L, Jing F, Jin H, Li T, Gu B, Wang L, Hao J, Zhao Y, Liu J, Zhang H, Li X, Li J, Ma W, Wang J, Normand ST, Herrin J, Armitage J, Krumholz HM, Zheng X; LIGHT Collaborative Group. Learning implementation of a guideline based decision support system to improve hypertension treatment in primary care in China: pragmatic cluster randomised controlled trial. BMJ. 2024 Jul 23;386:e079143. doi: 10.1136/bmj-2023-079143. PMID 39043397
- [Result] Chow CK, Klimis H, Thiagalingam A, Redfern J, Hillis GS, Brieger D, Atherton J, Bhindi R, Chew DP, Collins N, Andrew Fitzpatrick M, Juergens C, Kangaharan N, Maiorana A, McGrady M, Poulter R, Shetty P, Waites J, Hamilton Craig C, Thompson P, Stepien S, Von Huben A, Rodgers A; TEXTMEDS Investigators*. Text Messages to Improve Medication Adherence and Secondary Prevention After Acute Coronary Syndrome: The TEXTMEDS Randomized Clinical Trial. Circulation. 2022 May 10;145(19):1443-1455. doi: 10.1161/CIRCULATIONAHA.121.056161. Epub 2022 May 9. PMID 35533220
- [Result] Dorje T, Zhao G, Tso K, Wang J, Chen Y, Tsokey L, Tan BK, Scheer A, Jacques A, Li Z, Wang R, Chow CK, Ge J, Maiorana A. Smartphone and social media-based cardiac rehabilitation and secondary prevention in China (SMART-CR/SP): a parallel-group, single-blind, randomised controlled trial. Lancet Digit Health. 2019 Nov;1(7):e363-e374. doi: 10.1016/S2589-7500(19)30151-7. Epub 2019 Oct 10. PMID 33323210
- [Result] Schwarzbach CJ, Eichner FA, Rucker V, Hofmann AL, Keller M, Audebert HJ, von Bandemer S, Engelter ST, Geis D, Groschel K, Haeusler KG, Hamann GF, Meisel A, Sander D, Schutzmeier M, Veltkamp R, Heuschmann PU, Grau AJ; SANO study group. The structured ambulatory post-stroke care program for outpatient aftercare in patients with ischaemic stroke in Germany (SANO): an open-label, cluster-randomised controlled trial. Lancet Neurol. 2023 Sep;22(9):787-799. doi: 10.1016/S1474-4422(23)00216-8. Epub 2023 Jul 14. PMID 37459876